CLINICAL TRIAL: NCT04622059
Title: AUditive Direct In-utero Observation (AUDIO): Prenatal Testing of Congenital Hypoacusis
Acronym: AUDIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elena Contro (Other)
Responsible Party: Sponsor-Investigator, Elena Contro, consultant in fetal medicine, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Organization: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 104/2016/U/Sper
Record Dates: First submitted 2020-04-08; First posted 2020-11-09 (Actual); Last update posted 2021-03-18 (Actual); Status verified 2021-03

CONDITIONS: Hearing Loss
Keywords: RCT; prenatal testing of hypoacusis
MeSH Terms: conditions — Hearing Loss | interventions — Acoustic Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acoustic stimulation (Experimental): Fetuses in the group A (n=105) received an acoustic stimulation
  Interventions: Behavioral: acoustic stimulation
- no acoustic stimulation (No Intervention): Fetuses in the group B (n=105) no intervention was performed

INTERVENTIONS:
Behavioral: acoustic stimulation — An auditive stimulus was produced by hitting a diapason on an acoustic surface, at a distance of 2-3 cm from the mother's skin (in order to avoid mechanical vibration to reach the fetus) in the area near the fetus' head.
  The same procedure was repeated three times, waiting 30 seconds between one stimulus and the following one. The total duration of stimulation was about 2 minutes.
  Arms: acoustic stimulation

SUMMARY:
The objective of this randomized controlled study was to demonstrate whether fetal hearing can be assessed in utero.

DETAILED DESCRIPTION:
Unselected women at term of pregnancy (37-41 weeks of gestation) undergoing cardiotocography (CTG) according to routine clinical care and with a complete postnatal follow-up were consecutively recruited.

The two groups of women were selected in a random way, and it was an unblended randomization controlled trial (RCT), according to a list created by the website ww.randomization.com.

If the CTG was non-reactive for 10 minutes women who were eligible for the study were randomized into two groups.

An auditive stimulus was generated in group A. This stimulus was produced by hitting a diapason on an acoustic surface, at a distance of 2-3 cm from the mother's skin (in order to avoid mechanical vibration to reach the fetus) in the area near the fetus' head.

The same procedure was repeated three times, waiting 30 seconds between one stimulus and the following one. The total duration of stimulation was about 2 minutes. Cardiac accelerations on the CTG and fetal movements perceived by the mother were recorded in the ten minutes after the stimulus was produced.

No stimulation was produced in group B, but the CTG was prosecuted until the clinical criteria were satisfied. The total length of the CTG was variable from a minimum of 20 minutes to a maximum of one hour.

All the clinical variables were recorded in the Case Report Form (CRF) in particular the lapse of time needed for the first fetal cardiac acceleration and for the first fetal movement to occur.

A complete postnatal follow-up was obtained through the examination of medical records and parental interview.

A power analysis was carried out using Power Analysis Sample Size (PASS) software (Kaysville,UT,USA) and was conducted before the enrollment started. It was estimated that, for a survival comparison test (Log Rank), given the sample allocation ratio=1:1, 100 cases per group would be needed to validate a hazard ratio between group A and group B of 1.5 with a power of 80% and a Type I error of 5%.

ELIGIBILITY:
Inclusion Criteria:

1. Understand the Italian language;
2. Informative consensus;
3. To be between 18 and 48 years old;
4. To be sure of their gestational age, included between 37 0/0 and 41 5/7 weeks;
5. Single fetus pregnancy in cephalic position;
6. CTG with normal frequency and variability, without cardiac acceleration for 10 minutes, and with no uterine contractions.

Excluding criteria:

1. BMI before pregnancy more than 30 kg/m2, and at the end of pregnancy more than 35 kg/m2;
2. Uterine fibromatosis;
3. Premature rupture of membranes or oligohydramnios;
4. Fetal pathology (malformation or genetic syndromes);
5. Infective illness contract in pregnancy (CMV, herpes virus, rubella, syphilis, toxoplasmosis);
6. Anomalous CTG, or with contractions
7. Gestational diabet with insulin therapy;

7) Cholestasis of pregnancy; 8) Use of corticosteroids within the last hours; 9) Use of prostaglandins for cervical ripening, within the last hours.

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 210 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
First alteration of the CTG's reactivity | 40 minutes
  lapse of time between the acoustic stimulation and the alteration of the CTG's reactivity , the units of measure is minutes
First perception of fetal movements by the mother | 40 minutes
  lapse of time between the acoustic stimulation and the perception of fetal movements by the mother, the units of measure is minutes

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No